CLINICAL TRIAL: NCT02510976
Title: Prucalopride Versus Placebo in Functional Dyspepsia With Delayed Gastric Emptying
Brief Title: Prucalopride Versus Placebo in Gastroparesis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Prematurely stopped due to slow recruitment and expiry of study drug.
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S53094
Record Dates: First submitted 2015-07-27; First posted 2015-07-29 (Estimated); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis | interventions — prucalopride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prucalopride (Active Comparator): Prucalopride tablet 2 mg
  Interventions: Drug: prucalopride
- Placebo (Placebo Comparator): matching placebo tablet
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: prucalopride
  Other Names: Resolor
  Arms: Prucalopride
Drug: placebo
  Arms: Placebo

SUMMARY:
Controlled cross-over study of prucalopride 2 mg daily or placebo in gastroparesis (idiopathic or diabetic). Patients will be randomized to 4 week treatment with the first regimen (double-blind), followed by a 2-week washout and 4 week treatment with the second regimen in cross-over.

DETAILED DESCRIPTION:
To assess the influence of prucalopride (Resolor®) 2mg daily, 30 patients with idiopathic and 30 patients with diabetic gastroparesis will undergo two gastric emptying breath tests with concomitant assessment of meal-related symptoms, at the conclusion of two consecutive, 4-week treatment periods of prucalopride or placebo. The order of prucalopride and placebo treatment will be randomised at the initiation of the study. Medication for both patient groups, 30 patients with idiopathic and 30 patients with diabetic gastroparesis, will be randomized separately. Half of the subjects will receive placebo first; the other half will receive prucalopride first. Treatment periods will be separated by a wash-out period of 2 weeks. All drugs potentially affecting gastrointestinal motility or sensitivity will be discontinued at least two weeks prior to the initiation of the study. Informed consent will be obtained from each participant.

In order to establish the gastrointestinal symptom and quality-of-life profile of this cohort, each patient will complete the following validated self-reported instruments at baseline and at each of the two testing visits (table 1): Patients assessment of Gastrointestinal symptoms (PAGISYM), Patients assessment of Gastrointestinal Quality of Life Impact (PAGIQoL) Gastrointestinal and Global Severity Score, Patient Health Questionnaire (PHQ-15), Appetite Questionnaire, Hospital Anxiety and Depression Scale, Visceral Sensitivity Index, Short Form Nepean Dyspepsia Index (SF-NDI). The PAGI-SYM is a comprehensive questionnaire of upper GI symptoms, and it includes a gastroparesis questionnaire module: the Gastroparesis Cardinal Symptom Index (GCSI), which has been validated in (idiopathic) gastroparesis.26 Furthermore, during the entire study duration patients will complete a daily symptom diary, incorporating a separate horizontal 100-mm visual analogue scale (VAS) for each of 9 upper abdominal symptoms. As prucalopride has a well-known therapeutic effect in chronic constipation, patients will also register information about their stool frequency and stool type in the daily diary (Bristol Stool Scale).

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with a previously established diagnosis of diabetes or functional dyspepsia according to Rome III criteria, and with delayed gastric emptying (t1/2 for solids ≥ 109 min) on a breath test

Exclusion Criteria:

* The presence of oesophagitis, gastric atrophy or erosive gastroduodenal lesions on endoscopy

  * the presence of lesions on small bowel X-ray
  * major abdominal surgery
  * underlying psychiatric illness
  * use of non-steroidal anti-inflammatory drugs, steroids, or drugs affecting gastric motility.
  * Major co-morbidities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-11; Primary Completion 2021-01-08 (Actual); Study Completion 2021-01-08 (Actual)

PRIMARY OUTCOMES:
GCSI questionnaire score | after 4 weeks
  validated gastroparesis questionnaire

SECONDARY OUTCOMES:
PAGI SYM questionnaire scores | after 4 weeks
  validated upper GI questionnaire
NDI questionnaire scores | after 4 weeks
  validated upper GI QOL questionnaire
Gastric half emptying time | after 4 weeks
  gastric emptying test
Daily diary symptom and stool pattern scores | over 4 weeks, weekly average
  daily symptom diaries

OTHER OUTCOMES:
adverse events | over 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals, Leuven, Flanders, Belgium